CLINICAL TRIAL: NCT05699876
Title: A Comparative Study of Melatonin and Gabapentin as Premedication for Patients Undergoing Surgery Following Trauma
Brief Title: Melatonin vs Gabapentin for Post Trauma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kelika Prakash, Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIIMS Delhi
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Anxiety, Preoperarative
Keywords: melatonin; gabapentin; preoperative anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Melatonin; Gabapentin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental)
  Interventions: Drug: Melatonin 6 MG
- Gabapentin (Active Comparator)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Melatonin 6 MG — melatonin will be administered orally preoperatively as premedication
  Arms: Melatonin
Drug: Gabapentin — melatonin will be administered orally preoperatively as premedication
  Arms: Gabapentin

SUMMARY:
This project aims to compare the effect of preoperative administration of melatonin and gabapentin in reducing preoperative anxiety, stress markers and postoperative pain levels in trauma patients undergoing surgery. Gabapentin has analgesic as well as sedative properties. Melatonin, a hormone has been extensively used in intensive care units and has found to improve the sleep cycle and reduce pain. It is now being explored as a preoperative medication.

ELIGIBILITY:
Inclusion criteria: Patients will be recruited if they satisfy the following inclusion criteria:

* Age 18-65 years,
* ASA score I-II,
* Scheduled either for non-emergency surgery after trauma and
* Presumptive duration of operation not exceeding 3 hours.

Exclusion criteria: The following patients will be excluded from the study:

* Patients for emergency surgeries
* Surgeries taking place after 1pm (to account for diurnal variation in cortisol levels)
* Patients having altered mental state, history of psychiatric disorder, history of drug abuse or those on chronic pain medication
* Patients who have come for a repeat surgery and have already been included once in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
preoperative anxiety | 30 minutes after drug administration
  evaluate the difference in the preoperative anxiety score(Numerical Rating Scale ) before and after drug administration

SECONDARY OUTCOMES:
inflammatory markers | before and 30 minutes after drug administrartion
  o The serum cortisol and IL6 levels (biochemical markers of stress) intraoperatively and postoperatively
Sedation score | before and 30 minutes after drug administrartion
  Sedation score based on Observer Assessment of Alertness/Sedation Scale (OAA/S) before and after drug administration
post operative analgesia | 24 hours postoperative
  o Total fentanyl consumption 24 hours post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Aiims, New Delhi, National Capital Territory of Delhi, India